CLINICAL TRIAL: NCT06274528
Title: Effect of a Dual Orexin Receptor Antagonist on CSF Alzheimer's Disease Biomarkers
Brief Title: DORA and LP in Alzheimer's Disease Biomarkers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eisai Inc. (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Brendan Lucey, Professor of Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202301150; R01AG080551 (NIH)
Record Dates: First submitted 2024-01-29; First posted 2024-02-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
Keywords: Sleep; Older Adults; DORA
MeSH Terms: conditions — Alzheimer Disease | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lemborexant 10 mg (Experimental): Lemborexant is a capsule, taken by mouth once a night, approximately 30 minutes prior to bed for 6 months.
  Interventions: Drug: Lemborexant 10 mg
- Lemborexant 20 mg (Experimental): Lemborexant is a capsule, taken by mouth once a night, approximately 30 minutes prior to bed for 6 months.
  Interventions: Drug: Lemborexant 20mg
- Placebo (Placebo Comparator): Placebo is in capsule form and contains an inactive substance. It is taken by mouth once a night, approximately 30 minutes prior to bed for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant 10 mg — Within FDA approved dose 10 mg; capsule; QD, 6 month duration
  Other Names: DAYVIGO
  Arms: Lemborexant 10 mg
Drug: Lemborexant 20mg — 20 mg; capsule; QD; 6 month duration
  Other Names: DAYVIGO
  Arms: Lemborexant 20 mg
Drug: Placebo — 0 mg; capsule; QD; 6 month duration
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if the sleep aid, lemborexant, can decrease the amount of amyloid-beta and tau in the blood. Amyloid-beta and tau are proteins involved in the disease process leading to Alzheimer's disease.

DETAILED DESCRIPTION:
The overall goal of this project is to conduct an early stage (phase II) clinical trial of a dual orexin receptor antagonist (DORA), lemborexant, in cognitively normal older adults with amyloid deposition to demonstrate the feasibility and potential biological effectiveness of lemborexant's target engagement with multiple blood plasma and cerebrospinal fluid (CSF) Alzheimer's disease (AD) biomarkers. Orexins (also called hypocretins) are wake-promoting neuropeptides and blockade of orexin with a DORA increases sleep. The scientific premise of this project is that increased or enhanced sleep over 6 months by treatment with lemborexant will decrease the ratio of phosphorylated tau-181/tau-181 (pT181/T181) in blood and the concentration of CSF and plasma AD biomarkers (amyloid-β (Aβ), tau and phosphorylated tau (p-tau)) as well as neurodegeneration, inflammatory and synaptic AD biomarkers such as neurofilament light chain (NfL) (a non-tau marker of neuronal degeneration), soluble triggering receptor expressed on myeloid cells 2 (sTREM2) (a marker for immune response/microglial function), and neuronal pentraxin-2 (NPTX2) a marker for synaptic function) compared to placebo in amyloid-positive cognitively normal older adults. In addition, the investigators will also determine lemborexant's safety, pharmacokinetics (PK), and pharmacodynamics (PD) in this population. This study will enhance trial design and methods by providing critical information about dosing, safety, and target engagement of lemborexant on CSF and blood AD biomarkers to power phase III secondary prevention trials using lemborexant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Any race or ethnicity.
* Participants must be age ≥ 65 years and able to sign informed consent.
* Global Clinical Dementia Rating (CDR) 0.
* Willing and able to undergo study procedures.

Exclusion Criteria:

* History or reported symptoms suggestive of restless legs syndrome, narcolepsy, or parasomnia.
* STOP-Bang score >6 for participants without PAP.
* Untreated sleep apnea AHI>15
* Poorly treated sleep apnea due to noncompliance or an AHI ≥ 10.

  - PAP compliance is defined as ≥ 4 hours per night >70% of the nights.
* Plasma p-Tau217/np-Tau217% <2.5
* Stroke.
* History of renal impairment

  * Defined as older adult patients with markers of kidney damage or eGFR < 45.0 ml/min/1.73m2.
  * Normal Limits ≥ 45.0 mL/min/1.73m2
* History of hepatic impairment

  * AST and/or ALT ≥ 2X upper limit of normal (ULN).
  * Normal Limits: AST 11-47 IU/L and ALT 6-53 IU/L
* HIV/AIDS.
* History of substance abuse or alcohol abuse in the preceding 6 months.
* Regular alcohol consumption 3 or more days a week over the last 6 months. Regular alcohol consumption is defined as having more than 2 alcoholic beverages within 3 hours of bedtime. Participants that agree to reduce alcohol consumption during the study may not be excluded.
* History of presence of any clinically significant medical condition, behavioral or psychiatric disorder, or surgical history based on medical record or participant report that could affect the safety of the participant or interfere with study assessments or in the judgement of the Principal-Investigator (PI) if participant is not a good candidate.
* Has any medical condition that, in the PI's or study team investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the research procedures, or interfere with the collection/analysis of the data. Potential medical conditions that will be exclusionary at the PI's or study team investigator's discretion:

  * Cardiovascular disease requiring medication except for controlled hypertension.
  * Pulmonary disease.
  * Type I diabetes.
  * Neurologic or psychiatric disorder requiring medication.
  * Untreated depression
  * Tobacco use.
  * Use of sedating medications.
  * Use of medications that interact with lemborexant (if cannot be discontinued).
  * Abnormal safety labs.
* History of current suicidal ideations.
* Inability to speak and understand English.
* Currently pregnant or breast-feeding.
* In the opinion of the PI, the participant should be excluded due to an abnormal physical examination.
* Must not have participated in any clinical trial involving a study drug or device within the 30-days prior to study enrollment.
* Must not participate in another drug or device study prior to the end of this study participation.

Optional assessment exclusion criteria:

• Contraindication to lumbar puncture (anticoagulants; bleeding disorder; allergy to lidocaine or disinfectant; prior central nervous system or lower back surgery).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2029-03-11 (Estimated); Study Completion 2029-03-11 (Estimated)

PRIMARY OUTCOMES:
Changes plasma pT181/T181 ratio of lemborexant 10 and 20 mg compared to Placebo | 6 months
  plasma collection

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 6 months
  Adverse events
Measure the blood concentration of lemborexant 10 mg and 20 mg and determine the dose-response relationship with CSF pT181/T181 | 6 months
  Blood collection
Measure changes on blood plasma amyloid-beta isoforms (Aβ38, Aβ40, Aβ42, Aβ42/Aβ40) | 6 months
  Blood collection
Measure changes of CSF amyloid beta isoforms (Aβ38, Aβ40, Aβ42,Aβ42/Aβ40 ) | 6 months
  CSF collection
Measure changes of blood plasma p-tau/tau forms (T181, pT181, pT181/T181, S202, pS202, pS202/S202, T217, pT217, pT217/T217). | 6 months
  Blood collection
Measure changes of cerebrospinal fluid p-tau/tau forms (T181, pT181, S202, pS202, pS202/S202, T217, pT217, pT217/T217). | 6 months
  CSF collection

OTHER OUTCOMES:
Measure changes of cerebrospinal TREM2 (exploratory) | 6 months
  CSF
Measure changes of cerebrospinal NPTX2 (exploratory) | 6 months
  CSF
Measure changes of cerebrospinal NfL (exploratory) | 6 months
  CSF
Measure changes of blood plasma NfL (exploratory) | 6 months
  Blood

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lucey, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, School of Medicine, St Louis, Missouri, United States